CLINICAL TRIAL: NCT04009967
Title: Phase II Clinical and Translational Study of Neoadjuvant Pembrolizumab Before Radical Prostatectomy in Non-metastatic Gleason ≥8 Prostate Cancer Patients Positive by 18FDG-PET Scanning ( PICT-01)
Brief Title: Biomarkers for Neoadjuvant Pembrolizumab in Non-Metastatic Prostate Cancer Positive by 18FDG-PET Scanning
Acronym: PICT-01
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-910/OTSP-57
Record Dates: First submitted 2019-06-17; First posted 2019-07-08 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Pembrolizumab; 18FDG-PET Scanning
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prostate Cancer (Experimental): Participants will receive 3 cycles of pembrolizumab regardless of PD-L1 status. After completion of the second cycle of pembrolizumab treatment, and just before the third injection of pembrolizumab an 18FDG-PET/CT scan will be performed to assess a potential metabolic response. Then between 2 to 4 weeks after the third treatment, subjects will undergo radical prostatectomy. Subjects will be followed every 3 months during the first year post-surgery and according to physician decision during the following years.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg every three weeks for 3 cycles only
  Other Names: Keytruda

SUMMARY:
Various approaches are currently being developed for prostate cancer immunotherapy. However, a major challenge facing the development of cancer immunotherapy is the identification of tumors that would best respond to this type of treatment. Different studies suggest that prostate cancer more likely to progress are more infiltrated by exhausted T cells expressing the cell surface protein PD1 (Programmed cell death 1). Therefore, there is a strong rationale for selecting patients at higher risk of progression for testing the efficacy of anti-PD1 therapy.

High glucose metabolism as detected by fludeoxyglucose F18 (FDG)-positron emission tomography (PET) (18FDG-PET) imagery is an innovative biological biomarker-based method to identify patients at higher risk of recurrence and early failure to hormonotherapy. Recent study demonstrated that high intra-prostatic 18-FDG-uptake was associated with higher Gleason grades. Therefore the one third of Gleason ≥ 8 prostate cancer patients with higher 18FDG uptake would be ideal candidates for early immunotherapy treatments based on anti-PD-1 such as pembrolizumab.

The study aimed to identify biomarkers predictive the response to Pembrolizumab given prior to radical prostatectomy in participants with primary prostate cancer at high risk of progression.

DETAILED DESCRIPTION:
This is a Phase II, single-arm and open-label trial of pembrolizumab (MK-3475) in localized prostate cancer patients with newly diagnosed non-metastatic prostate cancer (Gleason grade ≥8 on biopsy) with positive tumor by FDG-PET (SUV max >4) who chose to undergo radical prostatectomy and lymph node dissection as primary treatment.

The trial will meet its endpoint if a reduction in cancer extent, proliferative index and increased apoptosis, as well as an induction of favorable immune cell infiltration and immune checkpoint expression profiles are observed after treatment compare to baseline..

ELIGIBILITY:
Inclusion Criteria:

* Male Age≥ 18 years old
* Non-metastatic prostate cancer with histologically confirmed Gleason sum ≥8
* Eligible for radical prostatectomy with a delay of 6 to 9 weeks
* Intraprostatic maximum standardized uptake value (SUVmax) ≥4 at 18-FDG-PET/CT exam.
* Not be castrated or under androgen deprivation therapy
* Not have received prior neo adjuvant hormonotherapy.
* Provided archival formalin-fixed, paraffin embedded tumor biopsy of the prostate tumor lesion not previously irradiated
* Performance status of Eastern Cooperative Oncology Group 0 to 1
* Adequate organ function

Exclusion Criteria:

* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4 (Cytotoxic T-lymphocyte-Associated Protein 4), OX-40, CD137).
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation.
* Has received prior radiotherapy to the prostate or other organs within 2 weeks of start of study treatment.
* Has received a live vaccine within 30 days prior to the first dose of study drug.
* Is participating or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Other primary cancer within 3 years
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has a known history of Hepatitis B or known active Hepatitis C virus infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is expecting to father children within the projected duration of the study, starting with the screening visit through the date of prostatectomy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
The antitumor activity of pembrolizumab assessed as the tumor response rate based on the change in tumor volume as measured by 18FDG-PET | Through study completion, an average of 1 year
  The change in tumor volume will be assessed by change in tumor volume from baseline after 3 cycles of pembrolizumab treatment
Mean difference change in proliferative index in prostate cancer patients between patients treated with pembrolizumab and the control cohort | Through study completion, an average of 1 year
  Proliferative index is measured by Ki67/apoptosis rate
Immune cell infiltration and immune checkpoint expression | Through study completion, an average of 1 year
  Compare large panel of ICP (Immune CheckPoints) ligand expression between patients treated by pembrolizumab and cohort control by imaging mass cytometry

SECONDARY OUTCOMES:
One year PSA (Prostate Specific Antigen) failure rate | At the end of study completion, an average of 3 years
  A statistically significant difference in the 1 year PSA failure rate compared to a historical cohort of untreated patients will indicate that the study has met this secondary objective.
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v4.0 | Through study completion, an average of 2 years
Number of participants with decrease in SUV uptake after 3 cycles of pembrolizumab | Through study completion, an average of 2 years
Assess a possible correlation between deficient mismatched repair (dMMR) and microsatellite instability-high (MSI-H) and response to pembrolizumab. | At the end of study completion, an average of 3 years
  dMMR and MSI-H status will be determined by immunochemistry and PCR (Polymerase Chain Reaction) respectively
Assess the expression of a series of cytokines and eicosanoids | At the end of study completion, an average of 3 years
  The concentration of 27 cytokines and 37 eicosanoids in tumor sample will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Yves Fradet, MD, Principal Investigator — CHU de Québec-Université Laval
Locations (1):
- CHU de Québec-Université Laval, Québec, Canada

IPD SHARING:
Plan to Share IPD: No